CLINICAL TRIAL: NCT04851860
Title: Effect of Sublingual Immunotherapy on Platlet factor4 Level in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Mohammad Mahmoud Mahmoud Elnaggar, Doctor Heba, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allergic rhintis in children
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Intervention Model Description: allergic rhintis children from 6 to12 years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allergic rhintis children (Other): sublingual immunotherapy is used for allergic rhintis children by dosing Allergen immunotherapy extract as sublingual drops which were kept under the tongue for a couple of minutes and then swallowed. The sublingual drops were administered in the morning on an empty stomach .
  Interventions: Drug: sublingual immunotherapy

INTERVENTIONS:
Drug: sublingual immunotherapy — sublingual immunotherapy is the only disease modifying therapy preventing the evolution of AR to asthma

SUMMARY:
Better management and improving outcome of children with allergic rhinitis

DETAILED DESCRIPTION:
The prevelance of Allergic Respiratory Diseases has been increased worldwide and affect 1of 5 persons of general population . ARDs are triggered by exposure to allergen and includes allergic rhinitis with or without conjunctivitis and bronchial asthma. ARDs are associated with decreased quality of life and increased economic burden .

Allergen-specific immunotherapy is the only disease modifying therapy preventing the evolution of AR to asthma, and its efficacy has long been known since observations by Leonard Noon in 1911. Allergen immunotherapy for AR is currently considered when showing strongly suggestive symptoms of AR which interfere with daily activities or sleep, and having evidence of IgE sensitization to ≥1 clinically relevant allergen .

The European Academy of Allergy and Clinical Immunology (EAACI) recommends treatmentof children with moderate to severe AR with Allergen Immunotherapy. It includes sublingual immunotherapy (SLIT) and subcutaneous immunotherapy (SCIT).Subcutaneous immunotherapy (SCIT) has been the gold standard, whereas sublingual immunotherapy (SLIT) has emerged as an effective and safe alternative .

Sublingual immunotherapy (SLIT) is the only treatment that regulates the immunological process during development of allergic rhinitis (AR), rather than simply treating symptoms.

Platelet activation occurs during antigen-induced airway reactions in allergic and asthmatic subjects. Raised levels of platelet-derived mediators, such as the Platelet Factor-4 (PF4), it is observed in plasma and bronchoalveolar lavage fluid of atopic individuals, and has the ability to activate eosinophils, increase expression of Fc-IgG and Fc-IgE receptors, and stimulate basophils to release histamine.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children with moderate to severe allergic rhinitis according to Allergic Rhinitis And Its Impact On Asthma (ARIA) guidelines[9], which interfere with daily activity or sleep.

  2. Children aged (6-12) years with clinical history of allergic rhinitis for at least one year.

  3. Children with allergic rhinitis who failed medical treatment, desire an alternative to pharmacotherapy.

  4. Sex : male and female.

Exclusion Criteria:

- 1. Children with chronic lung & heart diseases as: asthma and anatomical malformation for respiratory system.

2. disorders: Gastro Esophageal Reflux Disease, cystic fibrosis and epilepsy. 3.Children with chronic drug use: oral or nasal corticosteroids, antiepileptic and immunosuppressive.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-04-12 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
measurement of serum level of platlet factor 4 before and after sublingual immunotherapy | baseline
  diffrentiate serum level of platlet factor4 in children with allergic rhintis before and after treatment with sublingual immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Romeh, Study Director — Zagazig University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen Y, Zhou L, Yang Y. Effect of sublingual immunotherapy on platelet activity in children with allergic rhinitis. Braz J Otorhinolaryngol. 2017 Mar-Apr;83(2):190-194. doi: 10.1016/j.bjorl.2016.03.006. Epub 2016 Apr 22. PMID 27329923